CLINICAL TRIAL: NCT00319891
Title: Computer-Based Training for Mild Cognitive Impairment and Mild Alzheimer's Disease
Brief Title: Computer-Based Training for Mild Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUT-109-2005
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; AD; Mild Cognitive Impairment; Dementia; Cognitive remediation; computer-based training
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

INTERVENTIONS:
Procedure: Computer-based Cognitive Training

SUMMARY:
The primary objective of this study is to evaluate the effects of computer-based training program ("HiFi-AD") on the memory and cognitive abilities of individuals diagnosed with mild Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
The purpose of this study is to determine the extent to which computer-based cognitive remediation improves cognitive functions using standardized neuropsychological assessments relevant to AD; 2) the acceptability and feasibility of using computer-based cognitive remediation in an AD population.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English.
* Mini-Mental Status Examination (MMSE) score of 22 or higher.
* Adequate visual capacity.
* Adequate hearing capacity.
* Has a caregiver with some computer experience.
* Willing and able to commit to the time requirement of the entire study.

Exclusion Criteria:

* Clinically significant cerebrovascular disease.
* Participant is planning to begin acetylcholinesterase inhibitor (AChEI) therapy.
* Participants with severe tremor.
* Axis 1 or 2 psychiatric disorders.
* History of substance abuse.
* History of head trauma.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2004-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10

PRIMARY OUTCOMES:
The primary objective of this trial will be to assess the feasibility of using computer-based
cognitive training in an a population with early Alzheimer's Disease.

SECONDARY OUTCOMES:
A standardized set of neuropsychological assessments will be conducted pre- and post-
compuer-based training.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Kramer, PsyD, Principal Investigator — University of California, San Francisco; Kristine Yaffe, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States